CLINICAL TRIAL: NCT03604757
Title: Exploratory, Single-institution Study, Comparing 68Ga-RM2 PET/CT Versus 68Ga-PSMA-617 PET/CT in Patients Diagnosed With Prostate Cancer of Various Metastatic Risks Candidates for Radical Prostatectomy - "UROPET"
Brief Title: 68Ga-RM2 Compared to 68Ga-PSMA-617 PET/CT for Prostate Cancer Imaging According to Various Metastatic Risks
Acronym: UROPET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2016/38
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; 68Ga-RM2; bombesin; GRP-R; 68Ga-Prostate Specific Membrane Antigen; PSMA; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT Imaging (Experimental)
  Interventions: Drug: 68Ga-PSMA-617 PET/CT; Drug: 68Ga-RM2 PET/CT

INTERVENTIONS:
Drug: 68Ga-PSMA-617 PET/CT — PET/CT Imaging with 68Ga-PSMA-617 injection
Drug: 68Ga-RM2 PET/CT — PET/CT Imaging with 68Ga-RM2 injection

SUMMARY:
Patients with primary prostate cancer (low, intermediate or high metastatic risk) for whom radical prostatectomy is indicated, will be invited to participate to the present study.

Positron Emission Tomography coupled with scanner (PET-CT) using a radiotracer : 68Ga-RM2 and Positron Emission Tomography coupled with scanner (PET-CT) using another radiotracer : 68Ga-PSMA-617, will be scheduled.

DETAILED DESCRIPTION:
Approximately 15% of men with prostate cancer have high-risk disease at diagnosis. For these patients the accuracy of initial staging is of critical importance for treatment decision-making.

Recommended imaging modalities for initial staging include computerized tomography (CT) scan, bone scan, and Magnetic Resonance Imaging (MRI). In addition to initial work-up, 18F-Choline Positron Emission Tomography coupled with scanner (PET-CT) may be proposed in some high-risk patients but its sensitivity for lymph node detection remains limited.

Nowadays, new radiotracers are becoming available for prostate cancer imaging. Among them, PET-CT imaging with radiolabeled ligands of prostate specific membrane antigen (PSMA) could be more sensitive and more specific for the detection of lymph node metastasis in high-risk cancers, as it is the case with radiolabeled PSMA-617 which has demonstrated very promising results in men with metastatic prostate cancer in recent studies.

Therefore, PET imaging with 68Ga-PSMA-617 may participate to optimize work-up in the staging of high-risk patients.

Another family of radiopharmaceuticals aimed to target the Gastrin-Releasing Peptide Receptor (GRP-R) which is overexpressed in low-grade prostatic carcinomas. GRP-R expression is correlated with androgen receptor expression and with better outcomes.

Various radiolabeled GRP analogues have been developed and one of them, 68Ga-RM2, has shown very promising preclinical results. A study in 14 patients with prostate cancer showed encouraging results as related to the detection of primary prostate cancer and metastatic lymph nodes as well as in detection of local recurrence in the prostate bed and nodal relapse. However, 68Ga-RM2 failed to show some bone metastases in hormone-refractory patients. 68Ga-RM2 has also been recently used and compared to 68Ga-PSMA-11 for targeting biochemically recurrent prostate cancer. These radiotracers may offer complementary performances in lymph nodes detection due to their distinct pharmacokinetics.

Since 68Ga-RM2 and 68Ga-PSMA-617 target different cell populations, combining these two radiopharmaceuticals in patients could be of additional value.

The aim of this pilot study is to compare 68Ga-PSMA-617 PET/CT to 68Ga-RM2 PET/CT in 24 patients with prostate cancer of various progression risks to better understand how they could performed a metastatic risk mapping and how they could be used (or combined) in clinical practice.

ELIGIBILITY:
Inclusion criteria :

24 patients divided in :

* 6 patients with low risk prostate cancer (Gleason score ≤ 6 and cT1-T2a and Prostate Specific Antigen (PSA) value < 10 ng/mL)
* 12 patients with intermediate risk prostate cancer (Gleason score 7 or cT2b or PSA value 10-20 ng/mL) divided in : 6 patients who are Gleason score 7(3+4) (favourable intermediate risk) 6 patients who are Gleason score 7(4+3) (unfavourable intermediate risk)
* 6 patients with high risk prostate cancer (Gleason > 7 or cT2c or PSA value > 20 ng/mL)
* Candidate for radical prostatectomy after discussion in multidisciplinary committee
* Covered by the national health insurance system
* Written informed consent willingly obtained

Exclusion criteria :

* any kind of previous treatment for prostate cancer (hormonal treatment, EBRT, brachytherapy, cryotherapy, etc…);
* patient not candidate for radical prostatectomy and/or unable to benefit from surgery
* freedom deprivated patient by judiciary or administrative decision
* patient under legal protection or unable to express its own consent
* patient within exclusion period from another clinical trial
* known contraindication to radiopharmaceuticals and / or excipients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Median Standardized Uptake Value (SUV) | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
  Median Standardized Uptake Value (SUV) of 68Ga-PSMA-617
Median Standardized Uptake Value (SUV) | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
  Median Standardized Uptake Value (SUV) of 68Ga-RM2

SECONDARY OUTCOMES:
Gleason score | Day 3 to 60 (Last visit)
Receptor density Bmax | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
Local radioactive concentration (cpm) | Day 0 (inclusion) or Day 2 to 21 (Visit 2)
Immunoreactive score (IRS) | Day 3 to 60 (Last visit)

CONTACTS AND LOCATIONS:
Overall Officials: CLERMONT-GALLERANDE Henri, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No